CLINICAL TRIAL: NCT03541447
Title: A Pilot, Phase II Study With a Prospective, Randomized, Cross-Over, Placebo-Controlled, Double-Blind Design to Assess the Short-Term Effects of Tolvaptan Plus Placebo vs Tolvaptan Plus Octreotide LAR Combination Therapy in ADPKD Patients With Normal Kidney Function or Hyperfiltration
Brief Title: Tolvaptan-Octreotide LAR Combination in ADPKD
Acronym: TOOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Otsuka Pharmaceutical Italy S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOOL; 2017-004701-40 (EudraCT Number)
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD, Tolvaptan, Octrotide LAR
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tolvaptan plus Octreotide LAR / Tolvaptan plus Placebo (Experimental): Patients will receive a first 4-week treatment period with Tolvaptan up to 120 mg/die, according to tolerability, and a single dose of Octreotide LAR (two 20 mg i.m. injections). Then, after a period of wash-out, each patient will cross over to the other treatment arm for a second 4-week treatment period with Tolvaptan plus a single dose of placebo (two i.m. injections of 0.9% NaCl solution)
  Interventions: Drug: Tolvaptan; Drug: Octreotide LAR; Other: Placebo
- Tolvaptan plus placebo/Tolvaptan plus Octreotide LAR (Experimental): Patients will receive a first 4-week treatment period with Tolvaptan up to 120 mg/die, according to tolerability, and a single dose of placebo (two i.m. injections of 0.9% NaCl solution). Then, after a period of wash-out, each patient will cross over to the other treatment arm for a second 4-week treatment period with Tolvaptan plus a single dose of Octreotide LAR (two 20 mg i.m. injections).
  Interventions: Drug: Tolvaptan; Drug: Octreotide LAR; Other: Placebo

INTERVENTIONS:
Drug: Tolvaptan — Starting morning and afternoon doses of 45 and 15 mg, respectively, to be up titrated every two days to 60 and 30 mg and then to 90 and 30 mg, according to tolerability.
  Other Names: Jinarc
Drug: Octreotide LAR — A single dose of two 20 mg i.m. injections.
  Other Names: Sandostatin LAR
Other: Placebo — A single dose of two 20 mg i.m. injections.
  Other Names: NaCl 0.9%

SUMMARY:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is a leading cause of End Stage Kidney Disease (ESKD) worldwide. Elevated levels of 3', 5' - cyclic AMP (cAMP) play a central role in the pathogenesis and progression of the disease. Vasopressin antagonists and somatostatin analogues, which indirectly reduce adenyl cyclase 6 activity, have been found to markedly reduce renal tubular cell proliferation and cyst growth in experimental models of ADPKD. In combination, the two treatments show a clear additive effect and may significantly reduce renal cystic and fibrotic volume as well as cAMP levels to wild type levels.

The vasopressin antagonist Tolvaptan and the somatostatin analogue Octreotide share a similar renoprotective effect also in human disease.

Both medications effectively slow total kidney and cystic volume (TKV and TCV, respectively) growth and glomerular filtration rate (GFR) decline in patients with ADPKD. The short-term effect of both medications appear to be larger when the GFR is normal or even higher than normal and kidney volumes are still relatively stable. On the basis of experimental data, it is conceivable that Tolvaptan and Octreotide LAR should have an additive effect also in human disease, during initial treatment as well as in the long-term. To address the working hypothesis of an additional short-term effect of Tolvaptan and Octreotide, we propose to run a pilot, explorative, randomized, placebo-controlled, clinical trial with a Cross-Over Design to compare the short-term effects of Tolvaptan monotherapy and Tolvaptan plus Octreotide LAR combination therapy on TKV as assessed by MRI, and on GFR as directly measured by the iohexol plasma clearance technique in ADPKD patients with normal (80 to 120 ml/min/1.73m2) kidney function or even kidney hyperfiltration (GFR ≥120 ml/min/1.73m2).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18-yr-old) men and women, with a clinical and ultrasonographic diagnosis of ADPKD;
2. Serum creatinine < 1.0 mg/dl (for man) and < 1.2 mg/dl (for woman) and changes in serum creatinine (and creatinine clearance when available) <30% over the last six months;
3. Creatinine clearance > 80 ml/min/1.73m2 measured one to two weeks apart during the pre-screening period;
4. GFR ≥ 80 ml/min/1.73m2 (by iohexol plasma clearance technique) at screening and baseline evaluations;
5. TKV ranging between 1000 and 2000 ml at screening (by ultrasound imaging) and at baseline (by MRI) evaluations;
6. Female participants must be of non-childbearing potential or must agree to abstinence or use a highly effective form of contraception;
7. Written informed consent.

Exclusion Criteria:

1. Patients with concomitant systemic, renal parenchymal or urinary tract disease;
2. Diabetes;
3. Overt proteinuria (urinary protein excretion rate >1 g/24 hours);
4. Abnormal urinalysis suggestive of concomitant, clinically significant glomerular disease, urinary tract lithiasis, infection or obstruction, biliary tract lithiasis or obstruction;
5. Hemorrhagic or complicated cysts which might acutely affect kidney function and volumes;
6. QT-related ECG abnormalities;
7. Cancer and major systemic diseases that could prevent completion of the planned follow-up or interfere with data collection or interpretation;
8. Hypersensitivity to the IMP active substance or to any of the excipients or to benzazepine or benzazepine derivatives;
9. Concomitant treatment with drugs that may affect glomerular hemodynamics during the three months before the beginning of the study (including ACE inhibitors, angiotensin receptor blockers, aldosterone antagonists and non-steroideal anti-inflammatory medications);
10. Elevated liver enzymes and/or signs or symptoms of liver injury prior to initiation of treatment that meet the requirements for permanent discontinuation of tolvaptan
11. Patients with anuria, volume depletion and hypernatraemia
12. Patients who cannot perceive or respond to thirst
13. Ferro-magnetic prosthesis, aneurysm clips, severe claustrophobia or any other contraindication to MRI evaluation;
14. Psychiatric disorders and any condition that could prevent full comprehension of the purposes and risks of the study;
15. Pregnant or lactating;
16. Participation in another interventional clinical trial within the 4 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) | Changes from 4 weeks before randomization at baseline, 1,4,8,9,12 and 16 weeks after the randomization.
  GFR will be assessed by the Iohexol Plasma Clearance Technique

SECONDARY OUTCOMES:
Total Kidney Volume (TKV) | Changes from baseline at 4,8,12 and 16 weeks after the randomization.
  TKV will be assessed by Magnetic Resonance Imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — CRC per le Malattie Rare Aldo e Cele Daccò
Locations (1):
- CRC per le Malattie Rare Aldo e Cele Daccò, Ranica, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Trillini M, Caroli A, Perico N, Remuzzi A, Brambilla P, Villa G, Perna A, Peracchi T, Rubis N, Martinetti D, Caruso M, Leone VF, Cugini D, Carrara F, Remuzzi G, Ruggenenti P; TOOL Study Group. Effects of Octreotide-Long-Acting Release Added-on Tolvaptan in Patients with Autosomal Dominant Polycystic Kidney Disease: Pilot, Randomized, Placebo-Controlled, Cross-Over Trial. Clin J Am Soc Nephrol. 2023 Feb 1;18(2):223-233. doi: 10.2215/CJN.0000000000000049. PMID 36754009